CLINICAL TRIAL: NCT04580394
Title: Phase 2 Randomized Double-Blind Placebo-Controlled 4-Period Single-Dose Crossover Factorial Study to Evaluate the Contribution of the Individual Drug Components to the Efficacy of AD109 in Obstructive Sleep Apnea
Brief Title: Crossover Trial of AD109 in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-003
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AD109 (Experimental): Oral capsule administered before sleep
  Interventions: Drug: AD109; Diagnostic Test: Digit System Substitution Test
- Atomoxetine (Active Comparator): Oral capsule administered before sleep
  Interventions: Drug: Atomoxetine; Diagnostic Test: Digit System Substitution Test
- R-oxybutynin (Active Comparator): Oral capsule administered before sleep
  Interventions: Drug: R-oxybutynin; Diagnostic Test: Digit System Substitution Test
- Placebo (Placebo Comparator): Oral capsule administered before sleep
  Interventions: Drug: Placebo; Diagnostic Test: Digit System Substitution Test

INTERVENTIONS:
Drug: AD109 — Oral administration before bed
  Arms: AD109
Drug: Atomoxetine — Oral administration before bed
  Arms: Atomoxetine
Drug: R-oxybutynin — Oral administration before bed
  Arms: R-oxybutynin
Drug: Placebo — Oral administration before bed
  Arms: Placebo
Diagnostic Test: Digit System Substitution Test — a neuropsychological test sensitive to brain damage, dementia, age and depression where numbers are assigned symbols. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured.
  Other Names: DSST

SUMMARY:
This is a randomized, 4-period, placebo-controlled, crossover, phase 2 clinical study to examine the efficacy and safety of AD109 versus its individual components or placebo in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
The study is designed to examine the efficacy and safety of AD109 to treat obstructive sleep apnea. The study is a four-period single-dose randomized crossover design in which patients will undergo overnight polysomnographic (PSG) testing with dosing of one of the following 4 treatments: AD109, atomoxetine, R-oxybutynin or placebo. Participants will return 2 weeks after their final crossover PSG for an end of study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, between 25 to 65 years of age, inclusive, at the Screening Visit.
* AHI 10 to <20, or AHI ≥20 if meets other PSG criteria

Exclusion Criteria:

* History of narcolepsy.
* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control. A medication for these purposes is defined by dosage form, such that a combination antihypertensive medication is considered 1 medication
* CPAP should not be used for at least 2 weeks prior to first study PSG
* History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Empire Clinical Research, Pomona, California
  - Yale University, New Haven, Connecticut
  - Teradan Clinical Trials, Brandon, Florida
  - Clinical Trials of Florida, Miami, Florida
  - The Neurological Center of North Georgia, Gainesville, Georgia
  - CTI Clinical Research Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven clinical sites screened 146 participants, 60 participants were randomized. This was a double-blind, single dose crossover study. Participants underwent initial pre-screening to determine potential study eligibility. Overall study duration was up to 14 weeks. Participants who withdrew from the study were not replaced.
Pre-assignment Details: Participants underwent initial pre-screening to determine potential study eligibility. Patients selected for further screening had either a previous history of OSA of a severity consistent with enrollment criteria or had high risk.
Groups:
- All Participants: Oral capsules were administered before sleep in random order of each of the following: AD109 (Treatment A: Atomoxetine 75 mg and R-Oxbutynin 2.5 mg), Treatment B: Atomoxetine 75 mg and Placebo, Treatment C:R-Oxbutynin 2.5 mg and placebo, Treatment D:Placebo and Placebo. Each participant received single doses of each of the four treatments, the order in which each treatment was assigned was random.
Period: First Intervention
Arm/Group | All Participants
Started | 60
75mg/2.5mg (Treatment A: Atomoxetine 75 mg and R-oxybutynin 2.5 mg) | 16
75mg and Placebo (Treatment B: Atomoxetine 75 mg and placebo) | 14
2.5mg and Placebo (Treatment C: R-oxybutynin 2.5 mg and placebo) | 15
Placebo and Placebo (Treatment D) | 15
Completed | 57
Not Completed | 3
Not completed — Incorrectly Randomized | 1
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Period: Washout (One Week)
Arm/Group | All Participants
Started | 57
Completed | 56
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Second Intervention
Arm/Group | All Participants
Started | 56
75mg/2.5mg (Treatment A: Atomoxetine 75 mg and R-oxybutynin 2.5 mg) | 15
75mg and Placebo (Treatment B: Atomoxetine 75 mg and placebo) | 15
2.5mg and Placebo (Treatment C: R-oxybutynin 2.5 mg and placebo) | 13
Placebo and Placebo (Treatment D) | 14
Completed | 56
Not Completed | 0
Period: Washout (One Week)
Arm/Group | All Participants
Started | 56
Completed | 53
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Period: Third Intervention
Arm/Group | All Participants
Started | 53
75mg /2.5mg (Treatment A: Atomoxetine 75 mg and R-oxybutynin 2.5 mg) | 13
75mg and Placebo (Treatment B: Atomoxetine 75 mg and placebo) | 13
2.5mg and Placebo (Treatment C: R-oxybutynin 2.5 mg and placebo) | 15
Placebo and Placebo (Treatment D) | 14
Completed | 51
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Washout (One Week)
Arm/Group | All Participants
Started | 51
Completed | 49
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Fourth Intervention
Arm/Group | All Participants
Started | 49
75mg/2.5mg (Treatment A: Atomoxetine 75 mg and R-oxybutynin 2.5 mg) | 12
75mg and Placebo (Treatment B: Atomoxetine 75 mg and placebo) | 12
2.5mg and Placebo (Treatment C: R-oxybutynin 2.5 mg and placebo) | 11
Placebo and Placebo (Treatment D) | 14
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Oral capsule administered before sleep
  AD109 Atomoxetine R-Oxybutynin Placebo
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 47
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 33 [22 to 39]

OUTCOME MEASURES:

1. Primary Outcome: Change in Hypoxic Burden (HB) Log10HB[(%*Min)/Hour]
Description: Change in Hypoxic Burden (HB) is calculated as the oxygen desaturation 'area under the curve' in association with individual apneas and hypopneas. Due to the known logarithmic distribution of HB, data are primarily expressed and analyzed as Log10HB 4%[% min/hour]. Events with 4% or greater desaturations were included in the calculation of HB.
Time Frame: 1 night (treatment duration) (0-8 hours collected continuously)
Population: The efficacy was analyzed using the mITT Set comprised of all participants who took at least 1 dose of any of the study treatments and had at least 1 measurement for the primary endpoint. Fifty-nine (98.3%) participants were included in the mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Log10HB4%[%min/hour]
Arm/Group | AD109 | Atomoxetine | R-oxybutynin | Placebo
Number analyzed (Participants) | 59 | 59 | 59 | 59
Log10HB4%[%min/hour] | -0.41 [-0.54 to -0.28] | -0.36 [-0.49 to -0.23] | -0.04 [-0.17 to 0.09] | -0.06 [-0.18 to 0.07]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored for 14 weeks (Screening period, up to 4 weeks; 3-period crossover, up to 8 weeks; End of Study Evaluation, 2 weeks post crossover period).
Description: The study analysis did not analyze data by period. AEs were reported for the safety analysis by number and percent for treatment group only.
Groups:
- A: AD109: Treatment A: AD109 (Atomoxetine 75 mg + R-oxybutynin 2.5 mg)
- B: Atomoxetine 75 mg + Placebo: Treatment B: Atomoxetine 75 mg + Placebo
- C: R-oxybutynin 2.5 mg + Placebo: Treatment C:R-oxybutynin 2.5 mg + Placebo
- D:Placebo + Placebo: Treatment D: Placebo + Placebo
Arm/Group | A: AD109 | B: Atomoxetine 75 mg + Placebo | C: R-oxybutynin 2.5 mg + Placebo | D:Placebo + Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/54 | 0/54 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/54 | 0/54 | 0/57
Other Adverse Events (participants affected / at risk) | 2/56 | 2/54 | 0/54 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: AD109 (N=56) | B: Atomoxetine 75 mg + Placebo (N=54) | C: R-oxybutynin 2.5 mg + Placebo (N=54) | D:Placebo + Placebo (N=57)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pre-treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: AD109 (N=56) | B: Atomoxetine 75 mg + Placebo (N=54) | C: R-oxybutynin 2.5 mg + Placebo (N=54) | D:Placebo + Placebo (N=57)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agreed that because the Study is part of a Multi-center Study, individual publication could not be made until the publication of the Multi-center study results, notification that that a Multi-center publication was not planned, or after 18 months had passed

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT04580394/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04580394/SAP_001.pdf